CLINICAL TRIAL: NCT00385372
Title: Significance of an Elimination and Provocation Diet in Patients With Chronic Urticaria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Other Study IDs: BBU_PAD_CU_1
Record Dates: First submitted 2006-10-06; First posted 2006-10-09 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2007-02

CONDITIONS: Urticaria; Angioedema
Keywords: low pseudoallergen diet; elimination diet; provocation diet; oral provocation; natural food ingredients; food additives; flavours
MeSH Terms: conditions — Urticaria; Angioedema | interventions — Elimination Diets

INTERVENTIONS:
Procedure: elimination diet
Procedure: provocation diet

SUMMARY:
Patients with chronic urticaria undertake a five week elimination diet (pseudoallergen free diet). The efficacy of the diet will be determined by symptom score, by the use of rescue medication (oral antihistamines and glucocorticosteroids) and by a Quality of Life Questionnaire on week 0 and week 5. All patients with sufficient response (regarding the urticaria score) enter a second dietary part over six weeks, whereas a provocation diet is carried out. Each diet week a choice of pseudoallergen rich food is added, sorted by the type of pseudoallergens (e.g. biogenic amines, organic acids, flavours, additives). This study is conducted to investigate if the provocation diet could be a new diagnostic intervention to elucidate clinical relevant pseudoallergens.

DETAILED DESCRIPTION:
Chronic urticaria is defined as a daily or almost daily spontaneous occurrence of wheals that cause itching and lasting for at least six weeks. If there is no indication of a possible eliciting agent and because approximately 70% of patients benefit from it, a low-pseudoallergen diet should be carried out for 5 weeks. Although the low-pseudoallergen diet is successful, no explanation of the underlying mechanisms exists. On DBPC oral provocation testing with known food additives, only a small amount of patients, who experienced remission after a low-pseudoallergen diet react with new wheals and/or angioedema. For this discrepancy, natural food ingredients and new food additives are included in the dietary diagnostic. The high amount of substances, which are administrated within oral provocation testing can not reflect a realistic diet situation. Often it is impossible to ingest corresponding amounts of foods to reach the same concentration such as the provocation amount. Recording change reactions between food ingredients and the individual metabolism of the patients, the "step by step" food provocation method reveals itself to be most effective. In addition, individual predilections, amounts and frequency of ingested foods, are taken into consideration.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* chronic urticaria (duration: at least 6 weeks)
* patients who suffered from urticaria and/or angio oedema at least once a week for a duration of at least 4 weeks)
* Males and females, age between 7 and 80 years
* inpatients and outpatients
* oral antihistamines and glucocorticosteroids are allowed as concomitant medication (if needed)

Exclusion Criteria:

* pregnant or breastfeeding woman
* patients suffering from diabetes mellitus
* patients with cachexia
* known food allergies of food which will be administrated within the elimination diet (e.g. milk, cereals)
* isolated urticaria with known aetiology (e.g. physical urticaria, aquagene urticaria, urticaria factitia, cholinergic urticaria), Urticaria pigmentosa mastocytoses)
* patients, seemed to be uncompliant under suspicion of the investigator

Ages: 7 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 2005-01; Primary Completion 2007-01 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randolf Brehler, senior MD, Principal Investigator — University Hospital Münster, Department of Dermatology
Locations (1):
- University Clinics of Münster, Department of Dermatology, Münster, Germany

REFERENCES:
- [Result] Bunselmeyer B, Laubach HJ, Schiller M, Stanke M, Luger TA, Brehler R. Incremental build-up food challenge--a new diagnostic approach to evaluate pseudoallergic reactions in chronic urticaria: a pilot study: stepwise food challenge in chronic urticaria. Clin Exp Allergy. 2009 Jan;39(1):116-26. doi: 10.1111/j.1365-2222.2008.03110.x. PMID 19137651